CLINICAL TRIAL: NCT06450561
Title: Adherence to Secondary Prevention Guidelines for Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-60
Record Dates: First submitted 2024-06-03; First posted 2024-06-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Atherosclerosis; Stroke, Ischemic; Acute Coronary Syndrome; Ischemic Heart Disease; Peripheral Arterial Disease
MeSH Terms: conditions — Atherosclerosis; Ischemic Stroke; Acute Coronary Syndrome; Myocardial Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized due to a cardiovascular event: Patients hospitalized due to a cardiovascular event including stroke, acute coronary syndrome, ischemic heart disease, or peripheral arterial disease
  Interventions: Other: cardiovascular event

INTERVENTIONS:
Other: cardiovascular event — In this single group observational trial the exposure of interest is a cardiovascular event.

SUMMARY:
The present observational study aims to determine the degree of adherence to the recommendations of clinical guidelines regarding the prevention of cardiovascular complications in patients hospitalized due to a cardiovascular event.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the cardiology, neurology, or general surgery departments
* With any of the following admission diagnoses:

Non-ST-segment elevation acute coronary syndrome (NSTEACS) ST-segment elevation acute coronary syndrome (STEACS) Stable angina Unstable angina Non-ST-segment elevation myocardial infarction (NSTEMI) ST-segment elevation myocardial infarction (STEMI) Atherothrombotic ischemic stroke Lacunar stroke Peripheral artery disease Chronic ischemia of lower limbs Vascular ulcer due to arterial cause

Exclusion Criteria:

* Patients for whom lipid-lowering treatment is ruled out due to limited life expectancy
* Patients likely to die during hospitalization
* Patients who died during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized due to a cardiovascular event
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
patients admitted for a cardiovascular event who are prescribed lipid-lowering treatment at discharge | Up to 3 months
  Proportion of patients admitted for a cardiovascular event, warranting the initiation of secondary prevention with lipid-lowering agents, who are prescribed lipid-lowering treatment at discharge, adequate to reduce LDL by 50% or to below 55 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Tikhomirova, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari Alt Penedes i Garraf-Hospital Sant Camil, Sant Pere de Ribes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.